CLINICAL TRIAL: NCT05216367
Title: An Open-Label, Phase 1 Study to Assess the Effect of Hepatic Impairment on the Pharmacokinetics of Fruquintinib
Brief Title: Fruquintinib Hepatic Impairment Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2021-013-00US1
Record Dates: First submitted 2022-01-19; First posted 2022-01-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (healthy subjects) (Experimental): 8 healthy subjects with normal hepatic function will receive a single dose of 5 mg (1x5 mg) fruquintinib
  Interventions: Drug: Fruquintinib
- Cohort 2 (moderate hepatic impairment) (Experimental): 8 subjects with moderate hepatic impairment will receive a single dose of 2 mg (2 x 1 mg) fruquintinib
  Interventions: Drug: Fruquintinib
- Cohort 3 (mild hepatic impairment) (Experimental): 8 subjects with mild hepatic impairment will receive a single dose of 5 mg (1 x 5 mg) fruquintinib
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib will be administered as a single oral dose on the morning of day 1 under fasting conditions
  Other Names: HMPL-013

SUMMARY:
An Open-label, Phase 1 Study to Assess the Effect of Hepatic Impairment on the Pharmacokinetics of Fruquintinib

DETAILED DESCRIPTION:
This is a multicenter open-label, single-dose, single-period, sequential study in subjects without cancer with the primary objective of determining the effect of moderate and mild hepatic impairment on the PK of fruquintinib. The secondary objective is to evaluate the safety in subjects with moderate and mild (if enrolled) hepatic impairment and subjects with normal hepatic function.

Initially, subjects with moderate hepatic impairment will be enrolled. An interim pharmacokinetic (PK) analysis will be performed to evaluate the need to enroll subjects with mild hepatic impairment. Subjects with normal hepatic function will be enrolled after all other subjects have completed the study and will be matched for sex, age and body mass index. Subjects with hepatic impairment will be enrolled based on the hepatic function classification determined by Child-Pugh scoring.

Subjects with moderate hepatic impairment will receive a single dose of 2 mg fruquintinib to account for potential increase in fruquintinib PK exposure. Subjects with mild hepatic impairment or normal hepatic function will receive a single dose of 5 mg fruquintinib.

ELIGIBILITY:
Inclusion Criteria:

All Subjects

* Male or female between the ages of 18 and 75 years old (inclusive)
* BMI >18 and ≤40 kg/m2 and body weight not <50 kg at screening.
* Non-smoker or light smoker who smokes no more than 10 cigarettes, 2 cigars, 2 pipes, or other nicotine equivalents (eg, vape, snuff, gum) of tobacco per day; willing to limit smoking during the treatment period to 4 cigarettes or 1 cigar per day.
* Females must be of non-childbearing potential or surgically sterile
* Males who have not had a successful vasectomy and are partners of women of childbearing potential must use, or their partners must use, a medically acceptable method of contraception starting for at least 1 menstrual cycle prior to and throughout the entire study treatment phase, and for 2 weeks after the last dose of study drug. Those with partners using hormonal contraceptives must also use an additional approved method of contraception, such as a condom with spermicide. Males who have had a successful vasectomy (confirmed azoospermia, documentation needed) require no additional contraception.

Subjects with Hepatic Impairment

* For moderate hepatic impairment, the subject must have a Child-Pugh score of 7 to 9. For mild hepatic impairment, the subject must have a Child-Pugh score of 5 to 6
* The subject must have no clinically significant change in clinical condition within the last 30 days before screening
* The subject must have a condition consistent with hepatic impairment and associated symptoms but otherwise be determined to be in good health in the opinion of the Investigator.
* Subjects with ascites must not have a paracentesis within 3 months of screening.
* If diabetic, the subject must have the diabetes controlled (as determined by the Investigator).
* Concomitant medications to treat underlying disease states or medical conditions related to hepatic impairment are allowed. Subjects must be on a stable dose of medication and/or treatment regimen for at least 2 weeks before dosing as well as during the study.

Subjects with Normal Hepatic Function

* The subject must be without hepatic disease and have normal hepatic function
* The subject must be in good health

Exclusion Criteria:

All Subjects

* The subject has evidence of clinically significant cardiovascular, GI, renal, respiratory, endocrine, hematological, neurological, or psychiatric disease or abnormalities.
* The subject has a known history of any GI surgery or any condition possibly affecting drug absorption
* The subject has a clinically significant illness within 8 weeks or a clinically significant infection within 4 weeks prior to first dose
* The subject has a clinically significant ECG abnormality
* The subject has been diagnosed with acquired immune deficiency syndrome (AIDS) or tests positive for human immunodeficiency virus (HIV).
* The subject has clinically significant renal laboratory findings, including estimated creatinine clearance <60 mL/min as calculated by the Cockcroft-Gault equation.
* The subject has participated in a clinical study of another drug before screening, and the time since the last use of other study drug is less than 5 times the half-life or 4 weeks before day 1
* The subject has consumed grapefruit, starfruit, Seville oranges, or their products within 7 days prior to day 1.
* The subject has consumed herbal preparations/medications, including, but not limited to, kava, ephedra (ma huang), Ginkgo biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng, within 7 days prior to day 1.
* The subject has received blood or blood products within 8 weeks, or donated blood or blood products within 8 weeks prior to day 1 or donated double red cells within 16 weeks prior to day 1.
* The subject has experienced a weight loss or gain of >10% within 4 weeks prior to day 1 as documented by recent medical history and weight at screening to check-in (excluding subjects with moderate hepatic impairment).
* The subject has used any drug that is a strong inhibitor or inducer of CYP3A within 2 weeks (within 3 weeks for St. John's wort) prior to day 1 or will require use during the treatment period.
* The subject is allergic to the study drug or to any of its excipients.
* Female subject who is pregnant or planning to become pregnant, lactating, or breastfeeding.
* Male subject who plans to donate sperm or father a child within 3 months after receiving the study drug.

Subjects with Hepatic Impairment

* The subject has clinically significant vital sign abnormalities at screening or day -1
* The subject has used acetaminophen at doses >1 g/day within 2 weeks prior to study drug administration.
* The subject has a history or current diagnosis of uncontrolled or significant cardiac disease indicating significant risk of safety for participation in the study
* The subject has Gilbert's syndrome, liver transplant, Wilson's disease, autoimmune liver disease, esophageal variceal bleeding within 3 months prior to screening unless successfully treated with banding, known gastric varices, spontaneous bacterial peritonitis or paracentesis within 3 months before screening, cholestatic liver disease (eg, primary biliary cirrhosis or primary sclerosing cholangitis), history of biliary sepsis within the past 2 years, or a portosystemic shunt.
* The subject has previously diagnosed with hepatocellular carcinoma.
* The subject has acute or exacerbating hepatitis, fluctuating hepatic function, or rapidly deteriorating hepatic function as indicated by widely varying or worsening of clinical and/or laboratory signs of hepatic impairment in the judgment of either the Investigator or the Sponsor's medical monitor.
* The subject has a history of drug misuse within 6 months prior to screening or a positive drug test at screening or on day -1. A positive drug test may not be exclusionary if it is deemed to be the result of an approved prescribed concomitant medication.
* The subject has evidence of current or recent abuse of alcohol, which, in the Investigator's opinion, would compromise subject's safety or compliance with the study procedures or positive alcohol test at screening or on day -1
* The subject has received therapy known to exacerbate hepatic impairment within 2 weeks of day 1.
* The subject is taking antiviral therapy for treatment of active hepatitis infection at the time of screening.
* The subject has presence of clinically significant laboratory findings at screening are exclusionary, particularly:

  * Hemoglobin <8.5 g/dL
  * Platelet count <25,000/mm3
  * ALT or AST >5× upper limit of normal (ULN)
  * Hepatitis B surface antigen (HBsAg) positive and/or Hepatitis B core antibody positive
* The subject has systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg at screening or day -1

Subjects with Normal Hepatic Function

* The subject has evidence of clinically significant hepatic illness or abnormalities.
* The subject has evidence of a clinically significant deviation from normal in the physical examination, vital signs, or clinical laboratory determinations at screening or day -1
* The subject tests positive for Hepatitis B virus (HBV) assessed by the HBsAg and/or Hepatitis B core antibody, Hepatitis C virus (HCV), or Hepatitis C antibody.
* The subject has a history of drug or alcohol misuse within 6 months prior to screening or a positive drug test at screening or day -1
* The subject has used any prescription or non-prescription drugs, including over-the-counter (OTC) medications or vitamins, within 2 weeks prior to day
* The subject has systolic blood pressure >150 mmHg or diastolic blood pressure >95 mmHg at screening or day -1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
AUC 0-t | Day 1 to Day 11
  Area under the plasma concentration-time curve from time 0 to time of the last measurable concentration
AUC 0-inf | Day 1 to Day 11
  Area under the plasma concentration-time curve from time 0 to infinity (if data permit)
Maximum Plasma Concentration [Cmax] | Day 1 to Day 11
  To determine the maximum observed plasma concentration of Fruquintinib

SECONDARY OUTCOMES:
Incidence of Adverse Events/Serious Adverse Events | Day 1 to Day 11
  Any untoward medical occurrence associated with the use of study drug

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida